CLINICAL TRIAL: NCT05228353
Title: Clinical Audit of GI Endoscopic Complications in a Tertiary Care Hospital
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AIG/IEC-BH&R 14/05.2021-03
Record Dates: First submitted 2022-01-03; First posted 2022-02-08 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Endoscopy; Complication
Keywords: endoscopy; complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopy of the upper gastrointestinal tract using fiberoptic endoscopes was introduced in the late 1950s and provided the first opportunity for direct visualization of the esophagus, stomach, and duodenum and colon in vivo. GI Endoscopy is usually considered a safe and effective procedure. However complications do exist and procedure related costs are significant. There is a lack of prospective studies on complications of diagnostic and therapeutic endoscopic procedures.There is a lack of prospective studies on complications of diagnostic and therapeutic endoscopic procedures. Knowledge of potential endoscopic adverse events, their expected frequency, and the risk factors for their occurrence may help to minimize the incidence of adverse events. Review of adverse events as part of a continuing quality improvement process may serve to educate endoscopists, help to reduce the risk of future adverse events, and improve the overall quality of endoscopy.

DETAILED DESCRIPTION:
1. STUDY OBJECTIVES

1a. Primary objective - Clinical audit of complications in gastrointestinal endoscopy unit from a tertiary care centre.

1b. Secondary objective - NA

2. STUDY POPULATION- Consecutive patients coming to the hospital for any gastrointestinal endoscopic procedure for 6 months duration and develops a complication.

3. DESIGN AND DURATION OF THE STUDY- It will be an observational prospective audit of all consecutive patients coming to the hospital for any gastrointestinal endoscopic procedure for 6 months duration.

4. METHODOLOGY

4a. SUBJECT RECRUITMENT - All patients who undergo any diagnostic or therapeutic endoscopic procedure during the period and develop any complication.

4b. RANDOMIZATION AND BLINDING- N/A

4c. STUDY METHODS- This observational study will be conducted after obtaining ethical clearance from institutional human ethical committee. All patients who undergo any endoscopic procedure during the period including upper gastrointestinal endoscopy, colonoscopy, endoscopic retrograde cholangiopancreatography (ERCP), Endoscopic Ultrasound (EUS), Peroral Endoscopic Myotomy (POEM), Enteroscopy, Endoscopic mucosal resection (EMR), Endoscopic Submucosal Resection (ESD), Submucosal Tunnel Endoscopic Resection (STER), Anti Reflux Mucosal resection (ARMS), Anti Reflux Mucosal ablation (ARMA), GERD-X, Endoscopic Sleeve Gastrectomy (ESG) and develops an complication will be enrolled in the study.

4d. STUDY PROCEDURE- For each patient who develops a complication , Following variables will be collected: Details of procedure, Indication of procedure, H/O Antiplatelets, anticoagulants, Any co-morbidity, Operator Characteristics, Time of procedure, Duration of procedure, Type of sedation, Time of detection of complication, Length of hospital stay/ICU stay, Mortality, Financial Cost, 30 days Follow-up, Re-admission rate, American Society of Anaesthesiologists (ASA) physical status classification, Relevant Images of the procedure, Relevant Videos of the procedure.

4e. METHODS OF ASSESSMENT- As per clinical protocol, each patient will be assessed by the primary investigator at 24 hours after their procedure to assess for possible symptoms and complications and to answer any questions. Further, for the purposes of this study, all patients will be contacted by telephone 30 days or more after their procedure. A standardized telephone interview and a review of the electronic medical record will be used to obtain follow-up data. Following complications will be recorded as per ASGE guidelines.

1. Perforation
2. Bleeding
3. Infection
4. Pancreatitis
5. Cardio-pulmonary adverse event
6. Pain/ discomfort
7. Gas explosion
8. Thromboembolism
9. Instrumental penetration/ impaction
10. Drug reaction
11. Mortality

    4f.STOPPING OR DISCONTINUATION CRITERIA- N/A

    5. SAMPLE SIZE CALCULATION- Since this is a clinical audit, all the patients coming for GI endoscopic procedures and developing complications will be recorded.

    6. STATISTICAL ANALYSIS- Statistical analysis including both univariate and multivariate analysis, when appropriate, on available data. Univariate analysis will be conducted using chi-square test, Fisher's exact test, and relative risks with their 95% confidence intervals. Multivariate analysis of the main predictors of complications will be performed using a forward stepwise logistic regression model with the SAS statistical system. All candidate independent variables, age included, will be analyzed in a dichotomous manner.

    7. ETHICAL JUSTIFICATION OF THE STUDY- GI Endoscopy is a safe and effective procedure. However complications do exist and procedure related costs are significant. There is a lack of prospective studies on complications of diagnostic and therapeutic endoscopic procedures. This study aims to quantify and identify risk factors associated with endoscopy procedure complications. Knowledge of potential endoscopic adverse events, their expected frequency, and the risk factors for their occurrence may help to minimize the incidence of adverse events. Review of adverse events as part of a continuing quality improvement process may serve to educate endoscopists, help to reduce the risk of future adverse events, and improve the overall quality of endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo any diagnostic or therapeutic endoscopic procedure during the period and develop any complication including:

  * Diagnostic and therapeutic upper gastrointestinal endoscopy,
  * Diagnostic and therapeutic colonoscopy,
  * Endoscopic retrograde cholangiopancreatography (ERCP),
  * Endoscopic Ultrasound (EUS),
  * Peroral Endoscopic Myotomy (POEM),
  * Enteroscopy (Antegrade, Retrograde or spiral)
  * Endoscopic mucosal resection (EMR),
  * Endoscopic Submucosal Resection (ESD),
  * Submucosal Tunnel Endoscopic Resection (STER)
  * Anti- Reflex Mucosal Ablation (ARMA)
  * Anti- Reflex Mucosal Resection (ARMS)
  * GERD-X
  * Endoscopic Sleeve Gastrectomy (ESG)
  * Intra-gastric Balloon insertion

Exclusion Criteria:

* Those who are not willing to give the consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who undergo any diagnostic or therapeutic endoscopic procedure during the period and develop any complication will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42471 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical audit of GI Endoscopic complications in a Tertiary Care Hospital | 6 months
  The study aims to do audit of all endoscopic procedures occurring over six months duration and record any complications occurring during that period. Information related to the complications will be recorded.

SECONDARY OUTCOMES:
Risk factors for endoscopy complications | 6 months
  The information will be recorded to find risk factors for procedures so that future complication rate can be reduced. Besides this will help us in comparing the mortality and morbidity rate as compared with what is described in literature.
Morbidity associated with endoscopic complications | 6 months
  The study aims to review the morbidity associated with endoscopic complications during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Inavolu Pradev, MBBS, MD, DM, Principal Investigator — Consultant; Hardik Rughwani, MBBS, MD, DM, Principal Investigator — Consultant; Mohan ramchandani, MBBS, MD, DM, Study Director — Consultant; Nageshwar D Reddy, MBBS, MD, DM, Study Chair — Chief; Anudeep KV, MBBS, MD, DM, Principal Investigator — Consultant
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Result] Wolfsen HC, Hemminger LL, Achem SR, Loeb DS, Stark ME, Bouras EP, DeVault KR. Complications of endoscopy of the upper gastrointestinal tract: a single-center experience. Mayo Clin Proc. 2004 Oct;79(10):1264-7. doi: 10.4065/79.10.1264. PMID 15473407
- [Result] Mahnke D, Chen YK, Antillon MR, Brown WR, Mattison R, Shah RJ. A prospective study of complications of endoscopic retrograde cholangiopancreatography and endoscopic ultrasound in an ambulatory endoscopy center. Clin Gastroenterol Hepatol. 2006 Jul;4(7):924-30. doi: 10.1016/j.cgh.2006.04.006. Epub 2006 Jun 22. PMID 16797251
- [Result] Loperfido S, Angelini G, Benedetti G, Chilovi F, Costan F, De Berardinis F, De Bernardin M, Ederle A, Fina P, Fratton A. Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. Gastrointest Endosc. 1998 Jul;48(1):1-10. doi: 10.1016/s0016-5107(98)70121-x. PMID 9684657
- [Result] Levy I, Gralnek IM. Complications of diagnostic colonoscopy, upper endoscopy, and enteroscopy. Best Pract Res Clin Gastroenterol. 2016 Oct;30(5):705-718. doi: 10.1016/j.bpg.2016.09.005. Epub 2016 Sep 14. PMID 27931631
- [Result] Richter JM, Kelsey PB, Campbell EJ. Adverse Event and Complication Management in Gastrointestinal Endoscopy. Am J Gastroenterol. 2016 Mar;111(3):348-52. doi: 10.1038/ajg.2015.423. Epub 2016 Jan 12. PMID 26753887
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Derived] Katrevula A, Singla N, Rughwani H, Jagtap N, Katukuri GR, Godbole S, Teles de Campos S, Memon SF, Inavolu P, Singh AP, Mathur SS, Ashraf A, Patel R, Haja A, Asif S, Katamareddy T, Kalapala R, Ramchandani M, Lakhtakia S, Santosh D, Reddy N. Comprehensive audit of gastrointestinal endoscopy adverse events: Emphasizing quality indicators and economic impact with the AIG-AGREE modification. Endosc Int Open. 2024 Oct 28;12(10):E1242-E1250. doi: 10.1055/a-2435-5445. eCollection 2024 Oct. PMID 39474484